CLINICAL TRIAL: NCT04089683
Title: Evaluation of Bacterial Flora Among Operation Theatre Staff at a Tertiary Care Hospital - An Observational Prospective Study
Brief Title: Evaluation of Bacterial Flora Among Operation Theatre Staff at a Tertiary Care Hospital
Status: Completed | Type: Observational
Sponsor: Kamineni Academy of Medical Sciences and Research Centre (Other)
Responsible Party: Principal Investigator, Metta Jayachandra Reddy, Assistant Professor, Dept of Surgery, KAMSRC, Hyderabad, India, Kamineni Academy of Medical Sciences and Research Centre
Other Study IDs: KamineniAMSRC
Record Dates: First submitted 2019-09-06; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Microbial Colonization
Keywords: Operation Theatre; Bacterial Contamination; Web-space; OT Dress; Anterior Nares
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Doctors: Swabs collected from Web space, Scrub, Anterior nares before entering Operation theatre and while exit from operation theatre
  Interventions: Other: Swab stick
- Nurses: Swabs collected from Web space, Scrub, Anterior nares before entering Operation theatre and while exit from operation theatre
  Interventions: Other: Swab stick
- OT Technicians: Swabs collected from Web space, Scrub, Anterior nares before entering Operation theatre and while exit from operation theatre
  Interventions: Other: Swab stick
- House keeping staff and cleaners: Swabs collected from Web space, Scrub, Anterior nares before entering Operation theatre and while exit from operation theatre
  Interventions: Other: Swab stick

INTERVENTIONS:
Other: Swab stick — Swab sticks collected from Web Spaces, Scrub, Anterior Nares

SUMMARY:
Health care associated infection (HCAI) is a serious health hazard as it leads to increased morbidity and mortality of patients, length of hospital stay and costs associated with increased hospital stay.

A total of 361 subjects divided into four groups were included in this study. The first group comprised of 179 doctors, the second had 31 nurses, third group had 110 OT Technicians and the fourth group included 41 subjects which included housekeeping staff and cleaners. Swabs were collected from OT staff at the time of entry and at exit from the OT. Places of swabs taken were: A) Web space, B) OT dress and C) Anterior nares.

DETAILED DESCRIPTION:
Introduction:

Health care associated infection (HCAI) is a serious health hazard as it leads to increased morbidity and mortality of patients, length of hospital stay and costs associated with increased hospital stay. Infections from OT is well known and is well established which are often referred to as "hot zones" for emergence & spread of microbial resistance. Contamination in an operation theatre is an important cause of HCAIs and is the third leading cause of HCAIs.

This was a prospective observational study conducted in the operation theatre of a tertiary hospital once a month randomly from April 2014 - April 2016. All Operation theatre (OT) staff were included in the study. All the patients in OT and samples from the OT air & equipment were excluded from the study. A total of 361 subjects divided into four groups were included in this study. The first group comprised of 179 doctors, the second had 31 nurses, third group had 110 OT Technicians and the fourth group included 41 subjects which included housekeeping staff and cleaners. Swabs were collected from OT staff at the time of entry and at exit from the OT. Places of swabs taken were: A) Web space, B) OT dress and C) Anterior nares.

ELIGIBILITY:
Inclusion Criteria: All Operation Theatre staff -

Exclusion Criteria: Patients in Operation Theatre, Operating room air & equipment

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All OT staff viz. Surgeons, Anesthetists, Residents, OT matron/Nurse, OT Technicians, Housekeeping and Cleaning staff were include in the study. All the patients in OT and samples from the OT air & equipment were excluded from the study. All subjects were screened as per inclusion and exclusion criteria and selected without any gender bias.
  The study population contained 361 subjects among which were divided into four groups. Doctors, Nurses, OT technicians and others. Swabs were collected from OT staff at the time of entry in to OT and at the time of exit from OT. Places of swabs taken are: A) Web space, B) OT dress, C) Anterior nares (distal 1cm in a circular motion). Swabs were inoculated on 5% sheep blood agar/ Mueller-Hinton agar/ Mannitol salted agar/ MacConkey agar and were incubated at 35-37 degree centigrade under aerobic conditions for 48hrs with observation once in 24hrs. The age, gender and rank of the OT staff were collected as a part of demographic data.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Bacterial flora harboured at Web spaces among OT staff | 2 years
  Swabs will be taken from web spaces before entering Operation Theatre and while going out of OT at the end of the day and cultured to look for growth of Bacteria
Bacterial load on OT dress among OT staff | 2 years
  Swabs will be taken from OT dress while donning them and before going out of OT at the end of the day and cultured to look for growth
To identify the nasal carriers of organisms among OT staff | 2 years
  Swabs will be taken from anterior nares while entering OT at the end of the day while leaving OT and cultured to look for growth

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol